CLINICAL TRIAL: NCT05512039
Title: Reduced-dose onabotuLinumtoxinA for Urgency Incontinence Among Elder Females (RELIEF): A Randomized Controlled Comparative Effectiveness Trial With Embedded Qualitative and Costing Analyses
Brief Title: Reduced-dose Botox for Urgency Incontinence Among Elder Females
Acronym: RELIEF
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Dartmouth College (Other); University of Alabama at Birmingham (Other); University of Pittsburgh (Other); University of Texas (Other); Kaiser Permanente (Other); Oregon Health and Science University (Other); Stanford University (Other); University of Connecticut (Other); University of Nebraska (Other)
Responsible Party: Principal Investigator, Anne C. Cooper, MD MA, Principal Investigator, Assistant Professor, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY02001338
Record Dates: First submitted 2022-08-19; First posted 2022-08-23 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Overactive Bladder; Urinary Incontinence in Old Age; Urgency Urinary Incontinence
Keywords: Urinary Incontinence; Urgency Urinary Incontinence; Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Botox: Standard dose (Active Comparator): The standard dose of 100 units of botox will be injected into the bladder.
  Interventions: Drug: Botox 100 Unit Injection
- Botox: Low dose (Experimental): A lower dose of 50 units of botox will be injected into the bladder.
  Interventions: Drug: Botox 50 Unit Injection

INTERVENTIONS:
Drug: Botox 50 Unit Injection — Participants will be randomized to either receive a standard dose (100 units) or reduced dose (50 units) of onabotulinumtoxinA. If a participant has decreased symptom relief they may receive repeat treatment up to twice during the 12 month follow-up period, with minimum 4 month intervals between treatments.
  Other Names: OnabotulinumtoxinA 50 Unit Injection
  Arms: Botox: Low dose
Drug: Botox 100 Unit Injection — Participants will be randomized to either receive a standard dose (100 units) or reduced dose (50 units) of onabotulinumtoxinA. If a participant has decreased symptom relief they may receive repeat injection up to twice during the 12 month follow-up period, with minimum 4 month intervals between treatments.
  Other Names: OnabotulinumtoxinA 100 Unit
  Arms: Botox: Standard dose

SUMMARY:
The purpose of this study is to study the treatment of urgency urinary incontinence (UUI), specifically among women 70 years and older, by comparing reduced versus standard dose of onabotulinumtoxinA (BTX; trade name BOTOX(c)) injection in the bladder.

DETAILED DESCRIPTION:
The purpose of this quadruple-masked, randomized-controlled study is to study the treatment of urgency urinary incontinence (UUI) specifically among older women with low- versus standard-dose of onabotulinumtoxinA (BTX) via: symptom-specific and health-related quality of life (QOL; Aim 1), patient-reported and clinical outcome measures including adverse events (Aim 2), qualitative experience with focused interviews (Aim 3) and cost burden and economic impact (Aim 4). This study is an active collaboration between researchers in Gynecology, Urology, and Geriatrics at Dartmouth Hitchcock Medical Center (DHMC) and at 6 other centers; University of Alabama (UAB), University of Pittsburgh (U Pitt), University of Texas Southwestern (UTSW), Kaiser Permanente of Southern California (KPSCP), Oregon Health & Sciences University (OHSU), and University of Nebraska Medical Center (UNMC; joined January 2025). The investigators also have collaborators at Stanford University and University of Connecticut, though those sites are not recruiting participants.

ELIGIBILITY:
Inclusion Criteria:

1. Adult female at least 70 years old at date of enrollment
2. Urgency urinary incontinence (urge incontinence > stress incontinence per screening criteria)
3. On average 2 or more urgency or insensible incontinence episodes per day per patient report
4. Refractory urinary urgency incontinence, defined as

   1. Persistent symptoms despite trial of one or more conservative treatments (e.g. behavioral therapy, physical therapy, home Kegel exercises); participants not required to have attempted first line therapies if deemed not feasible or appropriate by provider with input of participant/caregiver.
   2. Persistent symptoms despite the use of anticholinergic and/or beta-3 agonist medication; or inability to tolerate medication due to side effects, or has a contraindication to taking medication, or is unable to afford the cost of the medication.
5. Currently not on an anticholinergic or beta-3 agonist medication or is willing to stop medication for 3 weeks prior to completing baseline bladder tally, with plan to remain off medication through duration of the study. Currently not actively using sacral neuromodulation therapy (either has not tried, or unit has been off for 4 weeks prior to baseline bladder tally and will remain turned off for the duration of the study). It is permissible for participants to continue self-led conservative therapies during participation in the study, including Kegel exercises, avoidance of bladder irritants, and urge suppression.
6. Willing and able to complete all study-related items, with assistance of caregiver(s) if needed.
7. Demonstrates awareness of possible need for catheterization in event of post-injection urinary retention & acknowledges risks of catheterization. Participant does not need to demonstrate ability to perform self-catheterization.
8. Grossly neurologically normal on exam and no gross systemic neurologic conditions believed to affect urinary function. Patients with a diagnosis of Parkinson's disease or diabetes may be eligible provided they have a grossly normal neurologic exam and otherwise fulfill the inclusion/exclusion criteria.

Exclusion Criteria:

1. Lack of capacity to provide consent. Will be assessed if needed per judgment of the site PI and study staff, with use of optional questionnaire.
2. Baseline persistently elevated post-void residual [PVR] (>150mL on 2 occasions in the 6 weeks prior to enrollment). If the PVR was obtained via bladder scanner with measurements differing by more than 100mL, or if there is concern about the accuracy of the scanner, it will be confirmed via catheterization which will be considered the gold standard.
3. Need for BTX injection to take place in the Operating Room or under sedation. (Of note, for repeat injection under the protocol, patients may have OR injection if indicated due to pain with initial BTX injection.)
4. Previous treatment with intravesical BTX in the last 12 months or use of sacral neuromodulation therapy within the past 4 weeks (unit may remain implanted, but should remain off for duration of the study).
5. Untreated symptomatic urinary tract infection (UTI). Eligible once UTI treatment complete and symptoms resolved.
6. Known bladder abnormality, including current or prior bladder malignancy, carcinoma in situ or untreatable cystitis (e.g. eosinophilic cystitis); prior major bladder surgery that would alter the detrusor muscle, such as augmentation cystoplasty; or hematuria that has not been evaluated.
7. Neurogenic detrusor overactivity or neurologic disease that may impact bladder function, including stroke, multiple sclerosis, peripheral neuropathy, spinal cord injury. Conditions such as Parkinson's disease and diabetes are acceptable provided normal bladder emptying and grossly normal neurologic function.
8. Concurrent BTX use for other indication, participants cannot exceed 300 units BTX in a 3 month period. Participants who may have conflict between study BTX administration and administration for other purposes may be excluded from participation if there is concern that study drug administration will be compromised. Concurrent use of BTX for another indication that would not exceed 300 units in a 3 month period, or that can have time of administration of the other BTX adjusted to avoid excessive dose, is acceptable; for instance, for migraines.
9. Greater than stage 2 pelvic floor prolapse, uncorrected or persistent despite pessary use (leading edge of prolapse not greater than 1cm beyond the hymen). Ongoing pessary use is permissible. Patients may have had a prior repair for pelvic organ prolapse. (see chart review of recent exam or perform brief exam while collecting post-void residual)
10. Planned prolapse or stress incontinence surgery; would defer enrollment to >3 months post-operative.
11. Allergy or intolerance to lidocaine or BTX.
12. Participation in another research study that could conflict with the RELIEF study, in estimation of the site PI.

Min Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 376 (Estimated)
Dates: Start 2023-05-12 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in symptom specific quality of life and bother over time. | Baseline, monthly post-injection through 12 months post-injection; primary outcome is at 3 months post-injection.
  The Overactive bladder questionnaire (OABq-SF), is a validated and reliable patient-centered quality of life questionnaire. The OABq-SF is based on a continuous sore of 0-100, with higher score translating to greater bother.

SECONDARY OUTCOMES:
Symptom severity | Baseline, 3, 6, & 12 months post injection. Results will be compared at the end of the 12 months.
  Urogenital Distress Inventory (UDI-6). The UDI-6 has a cut off score of 33.33 to distinguish women who are symptomatic versus asymptomatic. UDI-6 scores that are greater than 33.33 indicated higher distress caused by urinary incontinence symptoms.
Symptom bother | Baseline, 3, 6, & 12 months post injection. Results will be compared at the end of the 12 months.
  Incontinence impact questionnaire (IIQ). The IIQ has a cut off score of 9.52. This score distinguish women who are symptomatic and asymptomatic.
Change in number of urgency urinary incontinence (UUI) episodes per day. | Baseline, and 1, 3, and 6 months post injection
  Participants will keep a bladder tally for 3 days and results will be compared from baseline to 1, 3, and 6 months post injected to determine if there has been a change in the number of urgency urinary incontinence episodes.
Change in Global Symptom Improvement | Baseline,3, 6, & 12 months post injection
  Participants will be asked to complete the Patient Global Impression of Improvement (PGI-I) scale. The PGI-I scale is a one item assessment with responses ranging from "very much better" to "very much worse".
Goal setting and attainment | Baseline & 3 months post injection.
  Participants will express 3-5 goals and goal attainment will be assessed with the Patient Global Impression of Improvement Survey (PGI-I Scale). The PGI-I scale is a one item assessment with responses ranging from "very much better" to "very much worse".
Change in general health-related quality of life as measure by the Health Utility Index-3 | Baseline, 3 6 and 12 months
  Participants will complete the Health Utilities Index (HUI). The HUI measure health status, reporting health-related quality of life, and producing utility scores. The score ranges from 0.00 (dead) to 1.00 (perfect health).
Depression | Baseline, 3, 6 and 12 months post injection. Results will be compared at the end of the 3 month post injection.
  Patient Health Questionnaire-9 (PHQ-9) is a 10 item scale with scores ranging from 1(minimal depression) to 27 (severe depression).
Procedural discomfort and adverse events | Day of injection and monthly through 12 months
  Urinary retention, post-void residual & duration of voiding dysfunction; urinary tract infection, unscheduled clinic/emergency department visits and any adverse events assessed using the Clavien-Dindo scale,which has been validated for use in urology setting.
Qualitative experience of BTX treatment and adverse events | Baseline & 3 months post injection
  Using novel focused interview for a subset of participants. Participants will be interviewed before injection and 3 months post injection.
Survey of economic burden | Baseline, 3 & 12 months. Results will be compared at the end of the 12 months.
  Incontinence Resource Use Questionnaire measures the amount of use of various incontinence products. Questions include the number of incontinence protection items used per week.

CONTACTS AND LOCATIONS:
Overall Officials: Anne C Cooper, MD, MA, Principal Investigator — Dartmouth-Hitchcock Medical Center; E A Gormley, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (7):
- United States (7):
  - University of Alabama - Birmingham, Birmingham, Alabama
  - Kaiser Permanente Medical Group, San Diego, California
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Oregon Health & Science University, Portland, Oregon
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Yes, per PCORI data sharing policy. Details TBD.

REFERENCES:
- [Background] Amundsen CL, Komesu YM, Chermansky C, Gregory WT, Myers DL, Honeycutt EF, Vasavada SP, Nguyen JN, Wilson TS, Harvie HS, Wallace D; Pelvic Floor Disorders Network. Two-Year Outcomes of Sacral Neuromodulation Versus OnabotulinumtoxinA for Refractory Urgency Urinary Incontinence: A Randomized Trial. Eur Urol. 2018 Jul;74(1):66-73. doi: 10.1016/j.eururo.2018.02.011. Epub 2018 Feb 24. PMID 29482936
- [Background] Gormley EA, Lightner DJ, Faraday M, Vasavada SP; American Urological Association; Society of Urodynamics, Female Pelvic Medicine. Diagnosis and treatment of overactive bladder (non-neurogenic) in adults: AUA/SUFU guideline amendment. J Urol. 2015 May;193(5):1572-80. doi: 10.1016/j.juro.2015.01.087. Epub 2015 Jan 23. PMID 25623739
- [Background] Drake MJ, Nitti VW, Ginsberg DA, Brucker BM, Hepp Z, McCool R, Glanville JM, Fleetwood K, James D, Chapple CR. Comparative assessment of the efficacy of onabotulinumtoxinA and oral therapies (anticholinergics and mirabegron) for overactive bladder: a systematic review and network meta-analysis. BJU Int. 2017 Nov;120(5):611-622. doi: 10.1111/bju.13945. Epub 2017 Aug 2. PMID 28670786
- [Background] Coyne KS, Payne C, Bhattacharyya SK, Revicki DA, Thompson C, Corey R, Hunt TL. The impact of urinary urgency and frequency on health-related quality of life in overactive bladder: results from a national community survey. Value Health. 2004 Jul-Aug;7(4):455-63. doi: 10.1111/j.1524-4733.2004.74008.x. PMID 15449637
- [Background] Monz B, Pons ME, Hampel C, Hunskaar S, Quail D, Samsioe G, Sykes D, Wagg A, Papanicolaou S. Patient-reported impact of urinary incontinence--results from treatment seeking women in 14 European countries. Maturitas. 2005 Nov 30;52 Suppl 2:S24-34. doi: 10.1016/j.maturitas.2005.09.005. Epub 2005 Nov 16. PMID 16297579
- [Background] Furlong WJ, Feeny DH, Torrance GW, Barr RD. The Health Utilities Index (HUI) system for assessing health-related quality of life in clinical studies. Ann Med. 2001 Jul;33(5):375-84. doi: 10.3109/07853890109002092. PMID 11491197
- [Background] Horsman J, Furlong W, Feeny D, Torrance G. The Health Utilities Index (HUI): concepts, measurement properties and applications. Health Qual Life Outcomes. 2003 Oct 16;1:54. doi: 10.1186/1477-7525-1-54. PMID 14613568
- [Background] Yalcin I, Bump RC. Validation of two global impression questionnaires for incontinence. Am J Obstet Gynecol. 2003 Jul;189(1):98-101. doi: 10.1067/mob.2003.379. PMID 12861145